CLINICAL TRIAL: NCT02508896
Title: A Single-blind Phase 1 Study Assessing the Safety, Immunogenicity and Low Density Lipoprotein Cholesterol (LDLc)-Lowering Activity of 2 Different Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) Targeting AFFITOPE® Vaccines in Healthy Subjects
Brief Title: Study Assessing Safety, Immunogenicity and LDLc -Lowering Activity of 2 PCSK9 Targeting AFFITOPE Vaccines in Healthy Subjects
Acronym: AFF012
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Affiris AG (Industry)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AFFiRiS 012; 2015-001719-11 (EudraCT Number)
Record Dates: First submitted 2015-07-24; First posted 2015-07-27 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- AFFITOPE® AT04A+adjuvant (Experimental): 3 injections of 15µg AFFITOPE® AT04A+adjuvant once every 4 weeks and 1 boost immunization at a dose of 75μg, which will be applied one year after the 3rd immunization
  Interventions: Biological: AFFITOPE® AT04A+adjuvant
- AFFITOPE® AT06A+adjuvant (Experimental): 3 injections of 15µg AFFITOPE® AT06A+adjuvant once every 4 weeks and 1 boost immunization at a dose of 75μg, which will be applied one year after the 3rd immunization
  Interventions: Biological: AFFITOPE® AT06A+adjuvant
- Adjuvant without active component (Placebo Comparator): 3 injections of Placebo once every 4 weeks and 1 boost immunization which will be applied one year after the 3rd immunization
  Interventions: Biological: Adjuvant without active component

INTERVENTIONS:
Biological: AFFITOPE® AT04A+adjuvant — subcutaneous injection
  Arms: AFFITOPE® AT04A+adjuvant
Biological: AFFITOPE® AT06A+adjuvant — subcutaneous injection
  Arms: AFFITOPE® AT06A+adjuvant
Biological: Adjuvant without active component — subcutaneous injection
  Arms: Adjuvant without active component

SUMMARY:
Study AFF012 is a single blind, single-center, randomized, placebo-controlled, parallel group, phase I clinical trial of repeated administration by subcutaneous injection of a single dose of one of two different proprotein convertase subtilisin/kexin type 9 targeting AFFITOPE® vaccines or Placebo. This study will assess Safety, Immunogenicity and low density lipoprotein cholesterol-lowering activity of the two vaccines.

72 healthy subjects are divided into three test groups (2 treatment groups, 1 placebo group), each consisting of 24 subjects. The subjects are randomized to receive either of two AFFITOPEs® (AT04A or AT06A, adsorbed to 1 mg aluminium oxyhydroxide) or placebo (1 mg aluminium oxyhydroxide).

The study consists of 3 parts, part A, encompassing Visit 1 to Visit 8, covering 3 priming immunizations at a dose of 15μg at days 0, 28 and 56 and the immediate observation period extending to day 140; the prolonged observation period: part B, encompassing Visit 9 and Visit 10 at days 273 and 365; and part C consisting of 7 visits (V11 to V17). Study participants having received 3 priming vaccinations and having completed part B will receive in part C one boost immunization at a dose of 75μg, which will be applied one year after the 3rd immunization (day 420). Probands will proceed directly from part A to part B and to part C. Continuation of parts B and C will be considered based on the part A results, primarily the immunological results. The following scenarios apply (provided that there is no safety issue). None of the two treatment groups exhibits a vaccine-specific antibody response over the placebo group at Visit 8 - this will lead to termination of the trial. One of the two groups fails to exhibit a vaccine-specific antibody response over the placebo group at Visit 8 - this will lead to its discontinuation; the other treatment group and the placebo group will be continued.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 18 years of age at time of study entry.
2. Fasting LDLc at screening.
3. Fasting triglycerides at screening.
4. Body weight > 50 kg and a body mass index (BMI) between 19 and 35.

Exclusion Criteria:

1. Treatment/change in treatment with medications known to influence HDLc, LDLc and total cholesterol concentrations
2. Planned life-style changes during the study period like increasing aerobic exercise activity, attempting to lose body weight or changing the smoking status.
3. History of autoimmune diseases.
4. History of malignancy
5. Active or passive vaccination
6. Blood donation
7. History of severe hypersensitivity reactions and anaphylaxis.
8. History of allergic bronchial asthma.
9. Acquired or hereditary immunodeficiency.
10. Prior and/or current treatment with immune modulating drugs:
11. Subject has taken prescription lipid-regulating drugs
12. Treatment prior to screening with the following drugs: vitamin A derivatives and retinol derivatives for dermatologic treatment or any other drug known to influence cholesterol Levels
13. Infection with the human immunodeficiency Virus,Hepatitis B (HBsAg) or Hepatitis C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Occurence of any Serious Adverse Event (SAE) | 21 months
  Evaluation of SAE being unlikely, possibly, probably or definitely related to the study vaccines Occurence of any Grade 3 or higher adverse Event (AE) Occurence of solicited local AEs Occurence of solicited systemic AEs Occurence of unsolicited non-serious AEs

SECONDARY OUTCOMES:
Immunological activity of AFFITOPE® AT04A: Titer of vaccination-induced antibodies | 21 months
  Titer of vaccination-induced antibodies directed towards peptide components of the vaccine, the carrier, and the target proprotein convertase subtilisin/kexin type 9
Immunological activity of AFFITOPE® AT06A: Titer of vaccination-induced antibodies | 21 months
  Titer of vaccination-induced antibodies directed towards peptide components of the vaccine, the carrier, and the target proprotein convertase subtilisin/kexin type 9
Mean Levels of Low Density Lipoprotein Cholesterol (LDLc) | 21 months
  Change from baseline
Mean Levels of High Density Lipoprotein Cholesterol (HDLc) | 21 months
  Change from baseline
Mean Levels of Very Low Density Lipoprotein (VLDL) | 21 months
  Change from baseline
Mean Levels of Total Cholesterol (TC) | 21 months
  Change from baseline
Mean Levels of Triglycerides (TG) | 21 months
  Change from baseline
Mean Levels of PCSK9 | 21 months
  Change from baseline
Correlation analysis: Relating the strength of antibody responses to Lipid lowering effects | 21 months
  Relating the strength of antibody responses to Lipid lowering effects

CONTACTS AND LOCATIONS:
Overall Officials: Markus Zeitlinger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Zeitlinger M, Bauer M, Reindl-Schwaighofer R, Stoekenbroek RM, Lambert G, Berger-Sieczkowski E, Lagler H, Oesterreicher Z, Wulkersdorfer B, Luhrs P, Galabova G, Schwenke C, Mader RM, Medori R, Landlinger C, Kutzelnigg A, Staffler G. A phase I study assessing the safety, tolerability, immunogenicity, and low-density lipoprotein cholesterol-lowering activity of immunotherapeutics targeting PCSK9. Eur J Clin Pharmacol. 2021 Oct;77(10):1473-1484. doi: 10.1007/s00228-021-03149-2. Epub 2021 May 10. PMID 33969434